CLINICAL TRIAL: NCT06914531
Title: Assessment of the Development of Social Cognition in a Deaf Child With a Cochlear Implant : A Study Using a Standardized Questionnaire
Acronym: 1OL1
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/25/0073; ID-RCB : 2025-A00479-40 (Other: ANSM)
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Deaf Children; Cochlear Implant
Keywords: children; Cochlear Implants; Deafness; Social cognitive skills; Emotions skills
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- deaf child with a cochlear implant: This study focuses on children aged 3 to 6 years with congenital severe-to-profound deafness who received a cochlear implant before 15 months of age. The research aims to assess the adaptability of a standardized questionnaire evaluating social cognition in this population. Their communication abilities, response variability, and social interaction patterns are analyzed to refine assessment tools.
  Interventions: Other: Questionnaire comprehension test

INTERVENTIONS:
Other: Questionnaire comprehension test — Participants will complete a standardized questionnaire assessing social cognition, adapted for cochlear-implanted children aged 3 to 6 years. The assessment includes the Item Scale and the Test of Emotions Comprehension adapted and mixed together. The questionnaire evaluates children's ability to understand emotions, social interactions, and cognitive perspective-taking. Each child will complete the test in a single session lasting approximately 20 minutes, under the supervision of a trained investigator, with an orthophonist and a parent present

SUMMARY:
This study investigates the adaptability of a questionnaire assessing social cognition in children with cochlear implants aged 3 to 6 years, implanted before the age of 15 months. The primary objective is to evaluate the comprehensibility and relevance of the questionnaire in this population, considering their specific communication modes and cognitive profiles. By analysing response variability, communication abilities, and social interaction patterns, the study aims to refine the tool for accurate assessment. The findings will contribute to improving evaluation methods for social cognition in young deaf children.

DETAILED DESCRIPTION:
• Scientific Justification: Social cognition, particularly Theory of Mind, plays a crucial role in children's social interactions and emotional development. However, deaf children, especially those with cochlear implants, may experience delays or differences in Theory of Mind development due to limited access to spoken language and incidental learning. Assessing their social cognitive abilities requires tailored tools that accommodate their unique communication modes. This study aims to evaluate the adaptability and validity of a questionnaire designed to assess social cognition in deaf children aged 3 to 6 with cochlear implants. By analyzing communication strategies, response variability, and social interaction patterns, the research seeks to refine assessment methods, ensuring they accurately capture these children's cognitive and social competencies.

* The content of the responses: it is essential to measure this because it enables us to assess the quality of the children's reflections. Response content provides valuable insights into how deaf children with cochlear implants before 15 months perceive and interpret social interactions. This will allow us to test whether deaf children develop similar or different strategies for understanding the social world. Rich and relevant content would indicate good integration of social skills, which would be an indicator of success for the study.
* Understanding their own answers: it is important to check that the children understand what they are answering. This criterion is important because it ensures that the answers given are not the result of chance or a desirability bias, but of genuine reflection and a real understanding of social concepts. A child's understanding of his or her own responses is indicative of cognitive maturity and the ability to apply knowledge in social contexts, which is a central objective of the study.
* The degree of response, the completeness and accuracy of the answers given, is a key indicator of children's ability to understand and engage in cognitive tasks. This criterion measures the commitment and mental effort invested by the child in the exercise, as well as his or her ability to formulate detailed and relevant answers. A high level of response would be a positive sign of successful cochlear implantation in terms of cognitive and social development, while a low level of response could suggest difficulties in processing social information or expressing thoughts coherently.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 6 years old, who received a cochlear implant before the age of 15 months, who use their implant(s) and have a supportive family environment,
* Children with at least one cochlear implant undergoing speech therapy and are being monitored by the Pediatric Cochlear Implant Unit at Toulouse University Hospital,
* Children who are able to communicate: through speech, gestures, or French Sign Language,
* Children and their family whose mother tongue is French, - Social security coverage.

Exclusion Criteria:

* Cognitive or psychological impairment preventing the child from communicating,
* Other sensory or motor deficits that may interfere with pointing,
* Unstable psychiatric illness,
* Child whose parents both benefit from a legal protection measure.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consists of children aged 3 to 6 years with congenital severe-to-profound deafness who received a cochlear implant before 15 months of age.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2026-03-03 (Estimated); Study Completion 2026-03-03 (Estimated)

PRIMARY OUTCOMES:
Completion Rate of Standardized Social Cognition Questionnaire | Assessed during a single study visit (approximately 20-minute session).
  The primary outcome measure is the proportion of children who successfully complete all items of the standardized social cognition questionnaire. Success is determined by the child's ability to understand and respond coherently to the questions, demonstrating engagement and cognitive processing related to social interactions and emotions.

SECONDARY OUTCOMES:
Communication Ability During Questionnaire Completion | Assessed during a single study visit (approximately 20-minute session)
  Evaluation of the participant's ability to communicate while completing the questionnaire, including composite criterion with verbal, non-verbal (gestures, facial expressions), and mixed communication strategies. This will help assess whether children can effectively engage with the assessment.
Variability of Responses Among Participants | Assessed during a single study visit (approximately 20-minute session).
  Analysis of differences in questionnaire responses among participants. Variability will be examined based on factors such as age, duration of cochlear implant use, and language proficiency to determine individual differences in social cognition development.
Homogeneity of Responses Within the Study Group | Assessed during a single study visit (approximately 20-minute session).
  Assessment of response consistency across participants. Identifying patterns of similarity in answers will provide insight into shared cognitive and social processing abilities in cochlear-implanted children. High homogeneity could indicate a common understanding of the instructions and uniform accessibility of the questionnaire. Conversely, marked heterogeneity could reveal differences in the cognitive strategies used or in the interpretation of the items, requiring adaptation of the questionnaire.
Identification of Social Skills Demonstrated During the Assessment | Assessed during a single study visit (approximately 20-minute session).
  Observation and analysis of social behaviors exhibited by participants during the questionnaire session. This is a composite criterion who includes joint attention, emotional regulation, and perspective-taking, providing insight into their social cognitive abilities.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Toulouse - Pierre Paul Riquet, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fulcher A, Purcell AA, Baker E, Munro N. Listen up: children with early identified hearing loss achieve age-appropriate speech/language outcomes by 3 years-of-age. Int J Pediatr Otorhinolaryngol. 2012 Dec;76(12):1785-94. doi: 10.1016/j.ijporl.2012.09.001. Epub 2012 Oct 17. PMID 23084781
- [Background] De Giacomo A, Craig F, D'Elia A, Giagnotti F, Matera E, Quaranta N. Children with cochlear implants: cognitive skills, adaptive behaviors, social and emotional skills. Int J Pediatr Otorhinolaryngol. 2013 Dec;77(12):1975-9. doi: 10.1016/j.ijporl.2013.09.015. PMID 24466572
- [Background] Allen MC, Nikolopoulos TP, O'Donoghue GM. Speech intelligibility in children after cochlear implantation. Am J Otol. 1998 Nov;19(6):742-6. PMID 9831147